CLINICAL TRIAL: NCT00225394
Title: Long-Term Valcyte Therapy in Transplant Patients and the Development of Ganciclovir Resistant CMV
Brief Title: Long Term Use of Valganciclovir for Prophylaxis of CMV Disease in Kidney and Pancreas Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Lahey Clinic (Other); Rhode Island Hospital (Other)
Other Study IDs: VAL031
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2005-08

CONDITIONS: CMV Disease; Viral Resistance; Rejection; Death
Keywords: CMV; Kidney Transplant; Pancreas Transplant; Ganciclovir-resistance; Valganciclovir; CMV Disease
MeSH Terms: conditions — Rejection, Psychology; Death

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
CMV viral disease negatively affects transplant patients. CMV is the most prevalent infection in transplant patients and 3 month drug regimens to prevent the virus have been mostly unsuccessful, usually after the drug has been stopped, the patient develops the viral disease. Extended use of anti-viral drugs may, in fact, may lead to the development of resistant virus. We hypothesize that extended use (12 months) of valganciclovir (Valcyte™)will not only be efficacious but will not be associated with the development of resistant CMV.

Sample Size: 100 patients at 3 sites have been enrolled

Patient Selection: Adult (>18 years) recipients of cadaveric or living donor kidneys, pancreas, or combine kidney-pancreas transplants.

Immunosuppression: To be determined according to each center's standard protocol (s).

Study Drug: Valcyte™ Days 0 - 90: All Patients, 900 mg QD

Days 91 - 365:

Group 1: 900 mg QD Group 2: 450 mg QD

Assessment of Valgancicovir (Valcyte™)Resistant CMV : Serial serum samples (at transplant, 6 weeks, and 3, 6, 9 and 12 months post-transplant) for PCR amplification and DNA sequence analysis from detectable CMV to identify the presence of mutations within the UL97 and UL54 genes.

Other Analyses:

Additional information will be evaluated relating to the development of CMV disease, development of ganciclovir toxicity, graft rejection or graft loss and patient death. Preliminary information regarding the predictive value of DNA assays for the development of CMV disease will be evaluated.

DETAILED DESCRIPTION:
CMV infection occurs most frequently in the first three months following transplantation and following treatment for acute rejection; both instances can be related to relatively high levels of immunosuppression relative to stable long-term allograft recipients. Disease then can occur and is manifest as fever, low white blood cell count, pneumonitis, gastroenteritis, hepatitis, retinitis, and a multitude of other symptoms.

Ganciclovir, a potent inhibitor of the herpesviridae DNA polymerase encoded for on the unique long (UL54) region of the CMV genome, has had a significant impact on both the prophylaxis and treatment of CMV infection in transplant patients. CMV-infected cells produce a phosphotransferase, or kinase (UL97 region) that phosphorylates ganciclovir to ganciclovir-triphosphate. The triphosphate product inhibits CMV replication by competitively inhibiting the incorporation of deoxyguanine triphosphate (dGTP) into the DNA region encoding the polymerase (UL54 region), thus resulting in the premature termination of viral DNA synthesis. Resistance to ganciclovir is conferred when mutations occur on the UL97 region of the CMV genome.

Ganciclovir is available in either an oral or an intravenous formulation. The obvious advantages of the oral formulation are somewhat offset by the fact that its bioavailability is only 8 to 10%. The product has been reformulated with the addition of an L-valyl ester; the resulting compound, valganciclovir (Valcyte™) is metabolized to ganciclovir and has a 3 to 7 fold increase in bioavailability and is able to maintain serum concentrations equivalent to the intravenous formulation. This provides a convenient method for obtaining therapeutic concentrations of ganciclovir for extended periods of time without the need for in-dwelling intravenous lines.

The optimal length of treatment has not been established and relapse rates as high as 25% are common upon cessation of the antiviral agent.6 Patients with CMV disease are initially treated with intravenous ganciclovir for two or more weeks, and then with an oral agent for many weeks thereafter. Current laboratory technology allows detection of active viral replication, either through the detection of the pp65 antigen on the surface of infected leukocytes or through the use PCR amplification for the detection of viral DNA. It is however, still unclear whether the best therapeutic option is to treat until symptoms disappear or to treat until evidence of active viral replication ceases.

The question of whether or not prolonged exposure to ganciclovir will result in an increase in the incidence of resistant CMV strains has not been answered. There is also a theoretical increase in the risk of selection pressure for resistant CMV when the lower dose of valganciclovir (450 mg) is used. This proposal will document the emergence of ganciclovir-resistant strains of CMV in high-risk kidney, pancreas, or combined kidney/pancreas transplant patients receiving long-term suppressive therapy with Valcyte™ and will also address the issue of selection pressure by randomizing for low and high dose valganciclovir prophylaxis. Emergence of resistance will be defined as detection of a resistance-conferring mutation in the UL97 (phosphotransferase) or UL54 (DNA polymerase) open reading frame of detectable CMV.

Objectives

Primary

To document:

1. The emergence of ganciclovir-resistant CMV by PCR amplification and DNA sequence analysis for detecting resistance-conferring mutations of UL97 and/or UL54 open reading frames.
2. The development and time-to-onset of CMV disease

Secondary

To document:

1. The development of ganciclovir toxicity
2. Loss of kidney and/or pancreas graft function
3. Patient death

Tertiary

To attempt to determine the predictive value of DNA assays for the development of CMV disease.

Study Design

This will be a phase 4, 4 center, and randomized pilot study. Kidney, pancreas or combined kidney/pancreas transplant patients that receive induction anti-thymocyte globulin or OKT3 and/or are either seropositive for CMV or receive a graft from a CMV seropositive donor will receive Valcyte™ 900 mg daily for 90 days. Patients will then be randomized to either 450 mg or 900 mg Valcyte™ each day for days 91 to 365. Patients will be serially monitored for the development of ganciclovir-resistant CMV. Patients will receive standard immunosuppression, antibacterial and antifungal prophylaxis, and other necessary medications as determined by their physicians.

Statistical Analysis

Primary Endpoints: Time to development of any CMV disease or emergence of ganciclovir-resistant CMV.

Methods: Kaplan-Meier product limit estimates for median time to CMV disease for both treatment groups will be used, and a Kaplan-Meier survival curve will be plotted to compare treatment difference. Kaplan-Meier product limit estimates for median time to CMV resistance for both treatment groups will be used, and a Kaplan-Meier survival curve will be plotted to compare treatment difference. In addition, the Cox regression will be performed to compare treatment groups using treatment as a covariate in the model.

Secondary Endpoints: Incidence of ganciclovir toxicity, loss of kidney and/or pancreas, and patient death.

Methods: Cox regression will be performed to compare treatment groups using treatment and incidence of resistance as covariates in the model. Fisher's exact test will be used to analyze the loss of kidney and/or pancreas allograft function, and patient mortality. Toxicity within the two prophylaxis cohorts will be compared using Fisher's exact test, also.

Tertiary Endpoint: Efficacy of DNA assay to predict CMV disease. Method: A two-tailed t test comparison will be used to test the hypothesis that high copy numbers of CMV DNA correlate with the development of CMV disease. Additionally, a test based on a Cox proportional hazard model will be used to assess other variables and their impact on the development of CMV resistance and their relationship to copy numbers of DNA.

The above parameters will be assessed at three time points…6 months from the initiation of the trial, at 12 months post enrollment for each patient, and again at 24 months post-enrollment.

Materials and Methods

Definitions of CMV CMV Infection

CMV infection is defined as the isolation or identification of CMV from any site (blood, urine, sputum, stool), positive seroconversion (presence of positive CMV IgM or a four-fold increase in the titer of CMV IgG), or evidence of CMV viral replication (pp65 antigenemia or positive CMV by PCR amplification techniques) in the absence of clinical symptoms.

CMV Syndrome

CMV syndrome is defined as a virologically confirmed illness with any of the following: fever, pneumonia, leukopenia, lymphocytosis, thrombocytopenia, serum alanine aminotranferase levels > 2.5 x normal, with or without "flu-like" manifestations of viral immunity (malaise, myalgias, arthralgias, anorexia, nausea, vomiting). Any patient presenting with any of these signs or symptoms at any time during this study will have blood, body fluid, and/or biopsy specimen sent for viral confirmation which may include any of the following studies: histology for the presence of inclusion bodies, immunofluorescence of antibody to pp65 antigen or qualitative presence of CMV genome by PCR amplification.

CMV Disease

CMV disease will be defined as CMV infection and syndrome with any of the following: evidence of host cellular viral inclusions on biopsy or body fluid for cytology, a positive conventional viral culture for CMV, a positive "rapid antigen" test for the presence of pp65 antigen on the cell surface of buffy coat leukocytes, or the qualitative presence of CMV DNA as analyzed by PCR amplified virus. Specimens used for the above diagnostic procedures may include blood, liver or lung biopsy, endoscopic mucosal biopsy or brushing, bronchoalveolar lavage, or cerebrospinal fluid.

Severe CMV Disease

Severe CMV disease is defined as CMV disease in two or more organs or one or more of the following: CMV pneumonia, CMV retinitis, CMV CNS involvement, and invasive fungal or parasitic disease in association with CMV infection of any sort.

CMV Mortality

CMV mortality is defined as any death due to symptomatic CMV disease or death from any opportunistic infection while there is evidence of CMV disease or ongoing CMV viral replication.

Ganciclovir Resistant CMV

Ganciclovir resistant CMV is defined as the detection of a resistance-conferring mutation of the UL97 and/or the UL54 open reading frame by DNA sequence analysis of PCR amplified CMV genome.

Valganciclovir (Valcyte™)

Valcyte™ is a product of Roche Laboratories, Nutley, New Jersey. Patients will receive 450 or 900 mg per day depending on the stage of the study and the individual's randomization. Dosage will be adjusted for renal insufficiency as per package insert. If creatinine clearance (crcl) is >60 (ml/min), no adjustment is needed. If crcl is 40-59, patients can only receive up to 450 mg once daily. Therefore, those randomized to the 900mg/day cohort will receive 450 mg and those randomized to receive 450 mg/day will receive 450 mg every other day (QOD). If creatinine clearance is less than 40 and will never improve, patients will be excluded or terminated from the study.

Immunosuppression

Immunosuppressive medications will be administered according to the protocols in place at each participating center. The choice of maintenance immunosuppression and treatment for rejection will be at the discretion of the center's principal investigator.

Concomitant Anti-infectives

Patients enrolled in the study will receive anti-bacterial and anti-fungal prophylaxis as determined by the protocol in place for their transplanted organ at their transplant center. The use of antibiotics and anti-fungals for the treatment of disease will be at the discretion of the individual patient's physician.

Hematopoietic Growth Factors

Regrastim (GM-CSF) (Prokine® Hoechst-Roussel, and Leukine®, Immunex) and filgrastim (G-CSF) (Neupogen®, Amgen) may be used at the discretion of the physician for the treatment of leukopenia, including ganciclovir-related leukopenia.

ELIGIBILITY:
Inclusion Criteria:

1) Age greater than 18 years 2) WBC greater than 2000/mm3 with ANC greater than 500/mm3 3) Platelet count greater than 50,000/mm3 4) Hematocrit greater than 24 5) Life expectancy greater than 1 year as determined by investigator 6) Females must have a negative pregnancy test and any sexual partner must also agree to practice a barrier and/or hormonal method of birth control while participating in this study and for 90 days after. Females must agree to have a pregnancy test if a menstrual cycle is missed, and if positive, this must be reported.

-

Exclusion Criteria:

1. Patients receiving systemic therapy for acute opportunistic infection at time of enrollment
2. Patients receiving investigational drugs
3. Patients with malignancies within the last 5 years with the exception of excised basal or squamous cell skin cancers
4. Patients with active substance abuse or other condition that would impair compliance
5. Patients who are unable to give informed consent
6. Any patient with a creatinine clearance < 40 after delayed graft function and or post-transplant ATN has completely resolved, or the patient is deemed not to have the prospect of any further improvement of creatinine clearance (>40) as would occur with resolving ATN.
7. Persistent ANC < 1,000 for 2 consecutive weeks despite treatment with G-CSF
8. Any female patient who plans to become pregnant within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-10; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Uknis, MD, Principal Investigator — UMass Medical School
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Transplant, Burlington, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island